CLINICAL TRIAL: NCT06595017
Title: Evaluation of the Effect of Magnesium Sulfate Injection in Comparison to Lidocaine for Management of Myofascial Pain Dysfunction Syndrome: a Randomized Controlled Clinical Trial
Brief Title: Lidocaine Versus Magnesium Sulphate in Management of Myofascial Pain Dysfunction Syndrome
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Maha Abd ALMajied Mahmoud Mohamed, Demonstrator in Oral & Maxillofacial Surgery Department at Misr University for Science and Technology, Misr University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Myofascial Pain Dysfunction Syndrome
Keywords: Myofascial pain dysfunction syndrome; Magnesium Sulphate; Lidocaine; Pain; Electromyography
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Magnesium Sulfate; Lidocaine; Pharmaceutical Preparations; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Saline arm (Placebo Comparator): After localization of the trigger points, the skin was disinfected with alcohol, the tight muscle band was grabbed between two fingers, and a 30-gage 3/4-inch needle was introduced 1-2 cm away from the trigger points at a 30º angle to the skin. Negative aspiration was performed and each trigger point was injected with 2 ml of saline
  Interventions: Drug: Saline
- Lidocaine arm (Active Comparator): After localization of the trigger points, the skin was disinfected with alcohol, the tight muscle band was grabbed between two fingers, and a 30-gage 3/4-inch needle was introduced 1-2 cm away from the trigger points at a 30º angle to the skin. Negative aspiration was performed and each trigger point was injected with 2 ml of lidocaine
  Interventions: Drug: Lidocaine (drug)
- Magnesium Sulphate arm (Active Comparator)
  Interventions: Drug: Magnesium sulphate

INTERVENTIONS:
Drug: Magnesium sulphate — After localization of the trigger points, the skin was disinfected with alcohol, the tight muscle band was grabbed between two fingers, and a 30-gage 3/4-inch needle was introduced 1-2 cm away from the trigger points at a 30º angle to the skin. Negative aspiration was performed and each trigger point was injected with 2 ml of magnesium sulphate
  Arms: Magnesium Sulphate arm
Drug: Lidocaine (drug) — After localization of the trigger points, the skin was disinfected with alcohol, the tight muscle band was grabbed between two fingers, and a 30-gage 3/4-inch needle was introduced 1-2 cm away from the trigger point at a 30º angle to the skin. Negative aspiration was performed and each trigger point was injected with 2 ml of Lidocaine
  Arms: Lidocaine arm
Drug: Saline — After localization of the trigger points, the skin was disinfected with alcohol, the tight muscle band was grabbed between two fingers, and a 30-gage 3/4-inch needle was introduced 1-2 cm away from the trigger point at a 30º angle to the skin. Negative aspiration was performed and each trigger point was injected with 2 ml of Saline
  Arms: Saline arm

SUMMARY:
The goal of this clinical trial is to investigate the effectiveness of Magnesium Sulphate in the management of myofascial pain dysfunction syndrome in comparison to Lidocaine and Saline.

A total of 75 patients suffering from myofascial pain dysfunction syndrome will be assigned into one of three groups, each with 25 patients.

Group A: (Saline) includes patients enrolled for Saline injection into the trigger points. Group B: (Magnesium Sulphate) includes patients enrolled for Magnesium Sulphate injection into the trigger points. Group C: (Lidocaine) includes patients who will be enrolled for Lidocaine injection into the trigger points The primary outcome that will be investigated is (pain with a visual analogue score), and secondary outcomes will be (maximum mouth opening between edges of upper and lower incisors with millimeters, electrical activity with Electromyography, and quality of life assessed using the Oral Health Impact Profile questionnaire) The outcomes will be assessed pre-injection, 1month after injection, 3months after injection, and 6 months after injection

ELIGIBILITY:
Inclusion Criteria:

* Age Limitations: Participants must be between 18 and 55 years old.
* Chronic Pain Diagnosis: Individuals must have a diagnosis of chronic myofascial pain dysfunction syndrome (MPDS) affecting the face muscles, neck, shoulder, or upper back for a duration exceeding three months.
* Trigger Point Recognition: Patients must show awareness of their pain when pressure is applied to identified myofascial trigger points, in accordance with established diagnostic guidelines.
* Consent to Participate: Willingness to provide informed consent and engage in all aspects of the study.

Exclusion Criteria:

* Previous Treatments: A history of receiving dry needling or pulsed radiofrequency therapy, or currently participating in other pain management treatments.
* Recent Injury or Surgery: Any recent trauma, surgical procedures, or infections in the affected area within the past six months.
* Medication Interference: Current or recent use of moderate to strong analgesics (e.g., tramadol, morphine) that could influence pain assessment.
* Severe Health Conditions: Individuals with significant systemic illnesses (e.g., severe liver or kidney disease), blood clotting disorders, rheumatoid arthritis or epilepsy.
* Mental Health: Presence of current psychiatric disorders, cognitive impairments, or inability to comply with the study protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Pain score | At interval pre-injection and 1, 3, and 6 months after injection.
  Pain intensity was assessed using a 10-cm line visual analog scale (VAS) that represents a continuum between "no pain" and "worst pain." with 0 cm representing no pain, and 10 cm representing the worst pain imaginable.

SECONDARY OUTCOMES:
The maximum mouth opening | At interval pre-injection and 1, 3, and 6 months after injection.
  The maximum mouth opening (MMO) was evaluated by measuring the interincisal distance between the upper and lower central incisors.
Electrical activity | At interval pre-injection and 1, 3, and 6 months after injection.
  Measured using electromyography, EMG can provide valuable insights into altered muscle activity patterns and help in the diagnosis and management of myofascial pain dysfunction syndrome through readings.
Quality of life | At interval pre-injection and 1, 3, and 6 months after injection.
  evaluated using the Oral Health Impact Profile questionnaire (OHIP-14), which consists of 14 items categorized into seven domains of oral health. Participants were instructed to score each item on a scale from 0 to 4, where 0 indicates never, 1 represents hardly ever, 2 signifies occasionally, 3 denotes fairly often, and 4 corresponds to very often. The total score was computed by summing the responses to all 14 items, with higher scores reflecting a greater negative impact on oral health-related quality of life